## INFORMED CONSENT FORM (FOR INTERVENTION GROUP)

You have been invited to take part in a study titled 'The Effect of Nursing Care Based on Watson's Human Caring Model on the Quality of Life of Patients with Multiple Sclerosis'. This study is being conducted for research purposes. We recommend that you also participate in this study. Participation in the study is voluntary. Before deciding to participate in the study, it is important for you to know the purpose of the study and how it is being conducted, how your information will be used, and what the study includes. Please read the information below carefully and ask for clear answers to your questions. After you have been fully informed about the study and your questions have been answered, you will be asked to sign this form if you wish to participate.

What are the aims and basis of the study, and how many people other than me will participate in this study?

It was planned to evaluate the effect of nursing care based on Watson's Human Caring Model on the quality of life of patients. It is believed that the results of the study will guide nurses and other healthcare personnel working in this field. As a result of the literature review, there are very few studies in this field in our country regarding patients diagnosed with Multiple Sclerosis. It is thought that the study will contribute positively to patients and caregivers in this respect. 74 patients are expected to participate in this study.

• Should I participate in this study?

Whether or not you take part in this study is entirely up to you. If you decide to participate, this written informed consent form will be given to you to sign. Even if you sign this form now, you are free to leave the study at any time, without giving a reason. If you do not want to participate or leave the study, there will be no change in the treatment applied to you by your doctor. You also have the right to withdraw your consent at any stage of the study.

• What awaits me if I participate in this study?

In this study, you are first asked to fill out forms containing your introductory information and questions about your MS disease. In addition, we will complete our open-ended questions consisting of four questions by recording your voice with your permission. After the first interview, we will invite you to the hospital once a month for three months. In these interviews, we will provide you with training based on Watson's Theory of Human Caring. You will be asked to fill out the form again in the last week's interview. No risky situation or damage is foreseen in this research.

• What are the benefits of taking part in the study?

There is no medical benefit to you from the study. The aim is to improve your quality of life together with the nursing care you will receive. In addition, the results obtained from this study may be used for the benefit of other people. The study is for research purposes only.

What is the cost of participating in this study?

You will not be under any financial burden by participating in the study and you will not be paid anything.

• How will my personal information be used?

Your researcher will use your personal information to conduct the study and statistical analyses, and your identity will be kept confidential by your researcher throughout the study. At the end of the study, you have the right to request information about the results of the study. Information about

you cannot be viewed or disclosed by anyone else without your written permission. The study results may be used in scientific publications when the study is completed, but your identity will not be disclosed.

• Who can I contact for more information, assistance and contact?

If you have any problems with the study or need additional information about the study, you can reach Sevcan FİLİZ, who is conducting the study, at the phone number below.

Sevcan Filiz Mobile Phone Number: 0533 689 06 63

(Volunteer/Patient's Statement)

Specialist Nurse Sevcan FİLİZ stated that a medical study would be conducted and provided me with the above information about this study and I read the relevant text. After this information, I was invited to such a study as a "participant". I have understood all the explanations made to me in detail. Under these conditions, I agree to participate in the clinical study in question voluntarily, of my own free will, without any pressure or coercion.

- a. I have been informed that I have the right to refuse to participate in the study. I also know that this situation will not harm my medical care and my relationship with the physician.
- b. I am aware that I can withdraw from this study at any time without giving any reason, provided that I notify the responsible researcher. I understand that if I refuse to participate in this study or withdraw later, I will not be held responsible and that this will not affect the medical care I may need now or in the future in any way. (However, I am aware that it would be appropriate to notify the researchers in advance that I will withdraw from the study in order not to embarrass them.)
- c. The researcher who is the conductor of the study may remove me from the study without my consent, provided that my medical condition is not compromised by my negligence in fulfilling the requirements of the study program.
- d. The results of the study may be presented in scientific meetings or publications. However, in such cases, my identity will be kept strictly confidential.
- e. I do not assume any financial responsibility for the expenses incurred for the study. I will not be paid.

| Α | signed | copy o | of this | form | will b | oe : | given | to me. |
|----|--------|--------|---------|------|--------|----------|-------|--------|
| ٠. | 3.6 | cop, c | | | | <b>,</b> | D C. | |

date:

| Participant Name and Surname: |
|-------------------------------|
| Address: |
| Contact number: |
| signature: |